CLINICAL TRIAL: NCT06312345
Title: Ciprofol Versus Propofol for Anesthesia Induction in Cardiac Surgery: A Randomized Double-blind Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Le Yu (Other)
Responsible Party: Sponsor-Investigator, Le Yu, Clinicians, Shanghai East Hospital of Tongji University
Organization: Shanghai East Hospital of Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024.3.10-2024.5.1
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: ciprofol (Experimental)
  Interventions: Drug: Drug: ciprofol injection
- Placebo Comparator: propofol (Placebo Comparator)
  Interventions: Drug: Drug: ciprofol injection

INTERVENTIONS:
Drug: Drug: ciprofol injection — Patients in ciprofol group 0.3 mg/kg ciprofol for induction of anesthesia

SUMMARY:
Ciprofol, a novel intravenous general anesthetic with a chemical structure akin to propofol, boasts significantly enhanced potency. It offers a rapid onset, reduced incidence of injection pain, and minor impact on the cardiovascular system. However, clinical research regarding ciprofol's use for anesthesia induction in cardiac surgery remains limited.

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgery patients
2. Aged 55 to 75
3. New York Heart Association class II or III cardiac functions
4. Median sternotomy approach for coronary artery bypass grafting or heart valve replacement procedures

Exclusion Criteria:

1. With a history of benzodiazepine allergy
2. Significant liver or kidney insufficiency
3. Coagulation dysfunction
4. Neurological or psychiatric disorders
5. Undergone major surgery within the past three months.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-11 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | 1 second before induction of anesthesia (T1)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | 1 second before tracheal intubation (T2)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | 1 minute after tracheal intubation (T3)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | 5 minutes after tracheal intubation (T4)
  an average blood pressure in an individual during a single cardiac cycle
Heart beats | 1 second before induction of anesthesia (T1)
  the number of times each minute that heart beats
Heart beats | 1 second before tracheal intubation (T2)
  the number of times each minute that heart beats
Heart beats | 1 minute after tracheal intubation (T3)
  the number of times each minute that heart beats
Heart beats | 5 minutes after tracheal intubation (T4)
  the number of times each minute that heart beats

SECONDARY OUTCOMES:
Oxygenation index | 1 second before induction of anesthesia (T1)
  a calculation used in intensive care medicine to measure the fraction of inspired oxygen (FiO2) and its usage within the body.
Oxygenation index | 10 minutes after tracheal intubation (T5)
  a calculation used in intensive care medicine to measure the fraction of inspired oxygen (FiO2) and its usage within the body.
Injection pain | During procedure (When injecting the drug, ask the subject if the injection site is painful)
  Pain at the injection site when injecting the drug（Evaluation with Visual Analogue Scale）

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital of Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu L, Liu X, Zhao X, Shan X, Bischof E, Lu HH. Ciprofol versus propofol for anesthesia induction in cardiac surgery: a randomized double-blind controlled clinical trial. BMC Anesthesiol. 2024 Nov 12;24(1):412. doi: 10.1186/s12871-024-02795-0. PMID 39533186